CLINICAL TRIAL: NCT03605121
Title: Association Between Waist Circumference or BMI and Clinical Outcome in Cardiac Surgery
Brief Title: Waist Circumference in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, PhD, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: WC_cardiac surgery
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Abdominal
Keywords: waist circumference; body mass index; cardiac surgery; mortality
MeSH Terms: conditions — Obesity, Abdominal | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac surgery — The relationship between body mass index or waist circumference and clinical outcome in patients undergoing cardiac surgery will be assessed

SUMMARY:
Metabolic syndrome including increased body mass index or waist circumference is known to be a risk factor of cardiovascular disease. However, the relationship between body mass index or waist circumference and clinical outcome after cardiac surgery has not been fully elucidated.

DETAILED DESCRIPTION:
Along with body mass index, which is determined with height and weight, waist circumference reflects abdominal obesity and may increase cardio-metabolic risk and all-cause morbidity/mortality. In this observational study, we will review the electronic medical records of patients underwent cardiac surgery and assess their waist circumference, measured on preoperative computed tomography, as well as body mass index. The relationship between body mass index or waist circumference and mortality after cardiac surgery will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery between 2004 and 2016 at Seoul National University Hospital

Exclusion Criteria:

* Patients without information on height, weight, or waist circumference from abdominal computed tomography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery between 2004 and 2017 at Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
mortality | through study completion, average 3 years
  mortality after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided